CLINICAL TRIAL: NCT04872062
Title: Monitoring of Patients With Chronic Respiratory Failure Traeted With Non-invasive Home Ventilation: Contribution of New Monitoring Tools
Brief Title: Monitoring of Patients With Chronic Respiratory Failure Treated With Non-invasive Home Ventilation: Contribution of New Monitoring Tools
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, SOLER Julien, Hospital practitioner, Central Hospital, Nancy, France
Other Study IDs: 2020PI282
Record Dates: First submitted 2021-04-21; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Chronic Hypercapnic Respiratory Failure
Keywords: chronic hypercapnic respiratory failure; non-invasive ventilation; standardized NIV reading grid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic hypercapnic respiratory failure treated by home non-invasive ventilation (NIV)
  Interventions: Device: NIV cards; Other: Medical file

INTERVENTIONS:
Device: NIV cards — Reading the data available on the NIV cards
Other: Medical file — Using the data available in the medical file including clinical data, blood gas results, nocturnal oximetry results

SUMMARY:
Single-center retrospective study conducted on a population of patients with chronic hypercapnic respiratory failure treated by non-invasive ventilation at home, followed at the CHRU of Nancy. The objective is to assess the contribution of reading the NIV card with a standardized grid in their follow-up. The main objective is to assess the inter-observer agreement of a standardized NIV card reading grid, the secondary objective is to compare the results of NIV card reading between the usual NIV card reading method in the service and this same method completed by the addition of the standardized reading grid. The hypothesis is that the use of a standardized NIV card reading grid improves patient follow-up by standardizing their care.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Patients with chronic hypercapnic respiratory failure with a validated indication of long-term NIV
* Follow-up at the CHRU of Nancy at "Unité de Médecine Ambulatoire" (UMA) department between 11/01/2020 and 05/30/2021

Exclusion Criteria:

* Data not usable / missing
* Tracheal ventilation
* Patients' opposition to the use of their data for the purposes of this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic hypercapnic respiratory failure, treated with NIV at home, followed at the CHRU of Nancy in the UMA department between 11/01/2020 and 05/30/2021
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Agreement of responses to a standardized NIV reading grid between 2 observers | Day 0

SECONDARY OUTCOMES:
Comparison of the results between two observers between the method of reading NIV card usually performed in the department and this same method supplemented with a standardized NIV reading grid | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Julien Soler, Study Director — CentraHNF
Locations (1):
- CHRU de Nancy - Site de Brabois, Nancy, France